CLINICAL TRIAL: NCT06006338
Title: The Clinical Value of 3D Self-healing Elastic Liver Model for Surgical Training and Preoperative Planning: a Preliminary Study
Brief Title: 3D Printed Models for Liver Surgery
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Yuhua Zhang, MD, Vice director of Hepatobiliary and Pancreatic Surgery, Zhejiang Cancer Hospital, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: ZYH-CX-001
Record Dates: First submitted 2023-08-16; First posted 2023-08-23 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental)
  Interventions: Other: 3D Printed Model for preoperative planning

INTERVENTIONS:
Other: 3D Printed Model for preoperative planning — Besides conventional preoperative planning based on contrast-enhanced CT/MRI, the investigator refers to a 3D printed model to determine the optimal surgical approach via a trial-and-error method. Specifically, a personalized 3D printed model is fabricated. By referring to the printed model and CT/MRI images, a preliminary surgical trace is determined. Then, a simulation surgery is performed on the model, and surgical margin and the potential injury of vital vascular structures are evaluated. This assessment leads to the adjustment of the surgical path as necessary. The refined surgical route is then validated through a second simulation surgery performed on the healed 3D model. This iterative process is repeated multiple times, allowing for a comprehensive exploration of various approaches until the optimal surgical strategy crystallizes. Next, the investigator proceeds to execute the real surgery on the participant, meticulously adhering to the determined optimal surgical approach.

SUMMARY:
Comprehensive preoperative planning and real-time intraoperative guidance are essential prerequisites for achieving precise liver resection. In pursuit of this goal, the investigators have developed innovative 3D printed liver models utilizing a physically crosslinked self-healing elastomer created through the copolymerization of 4-acryloylmorpholine (ACMO) and methoxy poly (ethylene glycol) acrylate (mPEGA). These printed models exhibit exceptional healing capabilities, efficiently restoring their structure within minutes at room temperature, and rapidly recovering within moments after being incised.

Herein, the investigators aim to assess the viability of employing these 3D printed liver models as instrumental tools in designing the optimal surgical approach through an iterative trial-and-error methodology. Concurrently, the investigators aim to determine whether the integration of these 3D printed models into conventional methods (contrast-enhanced CT or MRI) can enhance the safety, ease, and efficiency of hepatic resection procedures.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years old;
2. Patients with a resectable tumor in the liver;
3. Eastern Cooperative Oncology Group Performance status score: 0;
4. Child-Pugh classification: A;
5. The Laboratory test results meet the following criteria and patients can tolerate surgery: Haemoglobin≥90g/L, Neutrophil count≥1.5×10⁹/L, Platelet count≥100×10⁹/L, Aspartate or alanine aminotransferase≤5 upper limits of normal(ULN）, alkaline phosphatase≤2.5 ULN, Serum albumin≥30g/L, serum creatinine<1.5 ULN, International normalized ratios（INR）≤2 or Prothrombin time（PT）exceed ULN≤6s, Creatinine clearance≥60 mL/min.

Exclusion Criteria:

1. Patients with extra-hepatic metastasis;
2. Anti-cancer therapy or surgery such as radiotherapy, radiofrequency ablation in 28 days prior to the surgery;
3. Clinically significant bleeding or bleeding tendencies within 3 months prior to enrollment or on thrombolytic or anticoagulant therapy;
4. Severe lung disease (eg, acute lung disease, pulmonary fibrosis that affects lung function, interstitial lung disease), uncontrolled diabetes mellitus (fasting blood glucose ≥10 mmol/L);
5. There are other unsuitable candidates for clinical trials, such as mental illness or alcohol dependence.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-02-29 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | 10 days
  The proportion of patients who achieved pathological negative surgical margin

SECONDARY OUTCOMES:
Injury of vital vascular structures | Immediately after the surgery.
  The Injury of vital vascular structures, such as portal veins or hepatic veins.
Operation time | Immediately after the surgery.
  Time length (minute) between the beginning and the end of the surgery.
Blood loss | Immediately after the surgery.
  The amount of lost blood (ml) in the operation.

CONTACTS AND LOCATIONS:
Overall Officials: Yuhua Zhang, Study Chair — Zhejiang Cancer Hospital
Locations (1):
- 1# Banshan East Rd. Zhejiang cancer hospital, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Lu Y, Chen X, Han F, Zhao Q, Xie T, Wu J, Zhang Y. 3D printing of self-healing personalized liver models for surgical training and preoperative planning. Nat Commun. 2023 Dec 19;14(1):8447. doi: 10.1038/s41467-023-44324-6. PMID 38114507